CLINICAL TRIAL: NCT01635660
Title: Prospective, Randomized, Multicentre Evaluation of Different Video-assisted, for Emergency Use Designed Intubation Aids for Out-of-hospital Endotracheal Intubation. Comparison of C-MAC System PM (Karl Storz), AP Advance (Venner Medical), and King Vision (King Systems) at Four German HEMS.
Brief Title: Out-of-Hospital Randomized Comparison of Video-assisted Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Karl Storz Endoscopy, Germany (Unknown); King Systems Corporation (Industry); LMA, Germany (Unknown); Venner Medical, Germany (Unknown)
Responsible Party: Principal Investigator, Erol Cavus, PD Dr. med. Erol Cavus, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANKIEL-VLS-2012-CAV
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Intubation Intratracheal; Airway Management; Emergency Treatment
Keywords: Out-of-hospital; airway management; intubation; video laryngoscope
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- C-MAC System (Active Comparator)
  Interventions: Device: Intubation
- AP Advance (Active Comparator)
  Interventions: Device: Intubation
- King Vision (Active Comparator)
  Interventions: Device: Intubation

INTERVENTIONS:
Device: Intubation — Tracheal Intubation with the assigned video laryngoscope

SUMMARY:
This research project examines the effectiveness of different video laryngoscopes in a out-of-hospital emergency intubation. Since in preclinical airway management severe incidents with esophageal failures of intubation may partly happen or rather endotracheal Intubation may completely fail, it is of great importance to evaluate alternative ways of endotracheal intubation in out-of-hospital emergency medicine. Video laryngoscopy has been proven in everyday clinical practice and may clinically be superior in most situations when compared to endotracheal Intubation using a conventional laryngoscope. No data exist, if different video laryngoscope types perform differently in the out-of-hospital setting. The investigators hypothesize that there would be no difference with regard to intubation time, intubation success, and intubation morbidity between different models of video laryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

- All adult emergency patients, age 18 years and older for whom a preclinical emergency intubation is necessary

Exclusion Criteria:

* Age under 18 years
* Laryngoscopy according to the algorithm of airway management not being indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Intubation success | Immediately after intubation

SECONDARY OUTCOMES:
Intubation on first attempt | Immediately after intubation
Intubation time | Immediately after intubation

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Klinikum LDW / NEF Bremen Süd, Bremen
  - Uniklinikum Greifswald / DRF Luftrettung, Greifswald
  - Uniklinikum Kiel / DRF Luftrettung, Rendsburg

REFERENCES:
- [Derived] Cavus E, Janssen S, Reifferscheid F, Caliebe A, Callies A, von der Heyden M, Knacke PG, Doerges V. Videolaryngoscopy for Physician-Based, Prehospital Emergency Intubation: A Prospective, Randomized, Multicenter Comparison of Different Blade Types Using A.P. Advance, C-MAC System, and KingVision. Anesth Analg. 2018 May;126(5):1565-1574. doi: 10.1213/ANE.0000000000002735. PMID 29239965